CLINICAL TRIAL: NCT03205293
Title: School-Based Intervention Program to Promote Healthy Eating and Physical Activity Using Participatory Approach
Brief Title: School-Based Intervention Program to Promote Healthy Eating and Physical Activity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Donna R Zwas, Director of Linda Joy Pollin Cardiovascular Wellness Center for Women, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2310SBI-HMO-CTIL
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Obesity, Childhood; Health Behavior; Physical Activity; Dietary Habits
Keywords: School-Based Intervention; Ecological Model; Participatory Approach; Palestinian Female Schoolchildren
MeSH Terms: conditions — Pediatric Obesity; Health Behavior; Motor Activity; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: This is a randomized control program trial, pre-post study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Female Schoolchildren, their mothers and teachers will be exposed to multiple interventions designed through a participatory approach, integrating the ecological model.
  Interventions: Behavioral: Intervention Program to Promote Healthy Eating and Physical Activity among Palestinian Female Schoolchildren
- Control Group (No Intervention): Regular school curriculum

INTERVENTIONS:
Behavioral: Intervention Program to Promote Healthy Eating and Physical Activity among Palestinian Female Schoolchildren
  Arms: Intervention Group

SUMMARY:
The purpose of this research is to develop, apply, and evaluate a school-based intervention program in East Jerusalem schools, designed to increase knowledge and to improve the attitudes and healthy behavior of schoolchildren, their teachers and their mothers' with regard to healthy eating and physical activity habits. The study tested the hypothesis that the impact of the entire school intervention program on students' lifestyles is mediated by their teachers' engagement in health promotion and by their mothers' involvement in school activity.

DETAILED DESCRIPTION:
A randomized controlled intervention program trial was carried out in 14 females' schools in East Jerusalem, selected randomly by a stratified sampling of four groups of schools. The primary target population was the students, while the secondary target populations were the mothers and the teachers at these schools. From the schools operating in East Jerusalem (Palestinian Authority, Jerusalem Municipality, private, and United Nations Relief and Works Agency) grades 4 and 5 were considered eligible to participate in the pre- and post-intervention studies.

The study process was designed, using the ecological model, in three stages; Stage one: Need assessment stage (pre-intervention, March-Jun 2011): A semi-structured interview was used with all 14 school principals, and a structured self-administered questionnaire was used with all teachers. A random sample of a 4th and 5th grade classes was selected, in which all mothers and their daughters were eligible to answer a self-administered questionnaire. The height and weight of the children were measured during this stage. These measurements were the baseline for assessing the current situation. In addition to school inspection tours was done to assess the school's health environment.

Stage two: Action stage (intervention, September 2011-June 2013): A random allocation of schools into intervention and control groups was done, followed by participatory planning and administration of the intervention in each of the 7 schools based on their needs assessments and assets. The program was implemented and administered by a steering committee in each of the schools, consisting of teachers, mothers, and children. Teachers underwent trainings in nutrition and physical activity. The program activities were monitored by regular visits twice a month. The implementation team met every four to six weeks to review the progress.

Stage three: Evaluation (post intervention, February-April 2013): Evaluation of the program was done after eighteen months of intervention using the same assessment questionnaires for both intervention and control schools among a different sample of children from grades 4 and 5, their mothers, and all of the teachers.

ELIGIBILITY:
Inclusion Criteria:

* East Jerusalem Female Schoolchildren

Exclusion Criteria:

* None

Ages: 4 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female Schoolchildren, their mothers and teachers
Enrollment: 1500 (Estimated)
Dates: Start 2011-03-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in percent of schoolchildren eating breakfast daily | At Baseline and 18 months after intervention
  Change in percent of schoolchildren eating breakfast will be assessed through a self report questionnaire based on the WHO's HBSC questionnaire
Change in percent of schoolchildren performing physical activity for ≥ 5 days per week | At Baseline and 18 months after intervention
  Change in percent of schoolchildren performing physical activity for ≥ 5 days per week will be assessed through a self report questionnaire based on the WHO's HBSC questionnaire
Change in percent of schoolchildren consuming the recommended servings of fruits and vegetables | At Baseline and 18 months after intervention
  Change in percent of schoolchildren consuming the recommended servings of fruits and vegetables will be assessed through a self report questionnaire based on the WHO's HBSC questionnaire
Change in teachers' engagement | At Baseline and 18 months after intervention
  Change in teachers' engagement will be assessed through a self report questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Donna Zwas, MD, MPH, Principal Investigator — Hadassah Medical Organization

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Diet, nutrition and the prevention of chronic diseases. World Health Organ Tech Rep Ser. 2003;916:i-viii, 1-149, backcover. PMID 12768890
- [Background] Wyatt SB, Winters KP, Dubbert PM. Overweight and obesity: prevalence, consequences, and causes of a growing public health problem. Am J Med Sci. 2006 Apr;331(4):166-74. doi: 10.1097/00000441-200604000-00002. PMID 16617231
- [Background] Lobstein T, Baur L, Uauy R; IASO International Obesity TaskForce. Obesity in children and young people: a crisis in public health. Obes Rev. 2004 May;5 Suppl 1:4-104. doi: 10.1111/j.1467-789X.2004.00133.x. No abstract available. PMID 15096099
- [Background] World Health Organization. The challenge of obesity in the WHO European Region and the strategies for response. Geneva: World Health Organization Regional Office for Europe, 2007.
- [Background] Badran M, Laher I. Obesity in arabic-speaking countries. J Obes. 2011;2011:686430. doi: 10.1155/2011/686430. Epub 2011 Nov 24. PMID 22175002
- [Background] Al Sabbah H, Vereecken C, Kolsteren P, Abdeen Z, Maes L. Food habits and physical activity patterns among Palestinian adolescents: findings from the national study of Palestinian schoolchildren (HBSC-WBG2004). Public Health Nutr. 2007 Jul;10(7):739-46. doi: 10.1017/S1368980007665501. Epub 2007 Feb 22. PMID 17381946
- [Background] Currie C, Hurrelmann K, Settertobulte W, Smith R TJ (editors). Health Behaviour in School-aged Children: a WHO Cross- National Study ( HBSC) International Report. Copenhagen: World Health Organization Regional Office for Europe; 2000.
- [Background] World Health Organization. WHO AnthroPlus for Personal Computers Manual. Geneva: World Health Organization, 2007.
- [Background] Mikki N, Abdul-Rahim HF, Shi Z, Holmboe-Ottesen G. Dietary habits of Palestinian adolescents and associated sociodemographic characteristics in Ramallah, Nablus and Hebron governorates. Public Health Nutr. 2010 Sep;13(9):1419-29. doi: 10.1017/S1368980010000662. Epub 2010 May 4. PMID 20441660
- [Background] Savige G, Macfarlane A, Ball K, Worsley A, Crawford D. Snacking behaviours of adolescents and their association with skipping meals. Int J Behav Nutr Phys Act. 2007 Sep 17;4:36. doi: 10.1186/1479-5868-4-36. PMID 17868479
- [Background] Alarcon de la Lastra C, Barranco MD, Motilva V, Herrerias JM. Mediterranean diet and health: biological importance of olive oil. Curr Pharm Des. 2001 Jul;7(10):933-50. doi: 10.2174/1381612013397654. PMID 11472248
- [Background] Guasch-Ferre M, Hu FB, Martinez-Gonzalez MA, Fito M, Bullo M, Estruch R, Ros E, Corella D, Recondo J, Gomez-Gracia E, Fiol M, Lapetra J, Serra-Majem L, Munoz MA, Pinto X, Lamuela-Raventos RM, Basora J, Buil-Cosiales P, Sorli JV, Ruiz-Gutierrez V, Martinez JA, Salas-Salvado J. Olive oil intake and risk of cardiovascular disease and mortality in the PREDIMED Study. BMC Med. 2014 May 13;12:78. doi: 10.1186/1741-7015-12-78. PMID 24886626
- [Background] Larson NI, Neumark-Sztainer D, Harnack L, Wall M, Story M, Eisenberg ME. Calcium and dairy intake: Longitudinal trends during the transition to young adulthood and correlates of calcium intake. J Nutr Educ Behav. 2009 Jul-Aug;41(4):254-60. doi: 10.1016/j.jneb.2008.05.001. PMID 19508930
- [Background] Dietary Guidelines for American 2005. U.S Department of Health and Human Services. Department of Agriculture. Available at: http://health.gov/dietaryguidelines/dga2005/document/pdf/dga2005.pdf (accessed: January 16, 2016).
- [Background] World Health Organization. Young People's Health in Context. Health Behaviour in School-aged Children (HBSC) Study: International Report from the 2001/2002 Survey. World Health Organization/ Europe. Available at: http://www.euro.who.int/en/publications/abstracts/young-peoples-health-in-context.- health-behaviour-in-school-aged-children-hbsc-study-international-report-from-the- 20012002-survey (accessed: January 18, 2016).
- [Background] Rolls BJ, Ello-Martin JA, Tohill BC. What can intervention studies tell us about the relationship between fruit and vegetable consumption and weight management? Nutr Rev. 2004 Jan;62(1):1-17. doi: 10.1111/j.1753-4887.2004.tb00001.x. PMID 14995052
- [Background] I.TETENS and S. ALINIA. The role of fruit consumption in the prevention of obesity. J Hortic Sci Biotechnol 2009;84:47-51.
- [Background] World Health Organization. Global Recommendations on Physical Activity for Health.Geneva : World Health Organization. Geneva, 2010. Available from: http://www.who.int/dietphysicalactivity/factsheet_recommendations/en/(accessed: February 11, 2016).
- [Background] American Academy of Pediatrics. Committee on Public Education. American Academy of Pediatrics: Children, adolescents, and television. Pediatrics. 2001 Feb;107(2):423-6. doi: 10.1542/peds.107.2.423. PMID 11158483
- [Background] Kanao BJ, Abu-Nada OS, Zabut BM. Nutritional status correlated with sociodemographic and economic factors among preparatory school-aged children in the Gaza Strip. J Public Health 2008;17:113-9.
- [Background] Jildeh C, Papandreou C, Abu Mourad T, Hatzis C, Kafatos A, Qasrawi R, Philalithis A, Abdeen Z. Assessing the nutritional status of Palestinian adolescents from East Jerusalem: a school-based study 2002-03. J Trop Pediatr. 2011 Feb;57(1):51-8. doi: 10.1093/tropej/fmq042. Epub 2010 Jul 31. PMID 20675716
- [Background] Temple JL, Giacomelli AM, Kent KM, Roemmich JN, Epstein LH. Television watching increases motivated responding for food and energy intake in children. Am J Clin Nutr. 2007 Feb;85(2):355-61. doi: 10.1093/ajcn/85.2.355. PMID 17284729
- [Background] Veldhuis L, Vogel I, Renders CM, van Rossem L, Oenema A, HiraSing RA, Raat H. Behavioral risk factors for overweight in early childhood; the 'Be active, eat right' study. Int J Behav Nutr Phys Act. 2012 Jun 15;9:74. doi: 10.1186/1479-5868-9-74. PMID 22704042
- [Background] Ouwens MA, Cebolla A, van Strien T. Eating style, television viewing and snacking in pre-adolescent children. Nutr Hosp. 2012 Jul-Aug;27(4):1072-8. doi: 10.3305/nh.2012.27.4.5805. PMID 23165544
- [Background] Pate RR, Mitchell JA, Byun W, Dowda M. Sedentary behaviour in youth. Br J Sports Med. 2011 Sep;45(11):906-13. doi: 10.1136/bjsports-2011-090192. PMID 21836174
- [Background] McDonald CM, Baylin A, Arsenault JE, Mora-Plazas M, Villamor E. Overweight is more prevalent than stunting and is associated with socioeconomic status, maternal obesity, and a snacking dietary pattern in school children from Bogota, Colombia. J Nutr. 2009 Feb;139(2):370-6. doi: 10.3945/jn.108.098111. Epub 2008 Dec 23. PMID 19106320
- [Background] Mirmiran P, Sherafat-Kazemzadeh R, Jalali-Farahani S, Azizi F. Childhood obesity in the Middle East: a review. East Mediterr Health J. 2010 Sep;16(9):1009-17. PMID 21218730
- [Background] Neuman M, Kawachi I, Gortmaker S, Subramanian SV. Urban-rural differences in BMI in low- and middle-income countries: the role of socioeconomic status. Am J Clin Nutr. 2013 Feb;97(2):428-36. doi: 10.3945/ajcn.112.045997. Epub 2013 Jan 2. PMID 23283503
- [Background] Doak CM, Visscher TL, Renders CM, Seidell JC. The prevention of overweight and obesity in children and adolescents: a review of interventions and programmes. Obes Rev. 2006 Feb;7(1):111-36. doi: 10.1111/j.1467-789X.2006.00234.x. PMID 16436107
- [Background] Hebert JR, Clemow L, Pbert L, Ockene IS, Ockene JK. Social desirability bias in dietary self-report may compromise the validity of dietary intake measures. Int J Epidemiol. 1995 Apr;24(2):389-98. doi: 10.1093/ije/24.2.389. PMID 7635601